CLINICAL TRIAL: NCT02692326
Title: DECREASE OF CHOLESTASIS USING CYCLED PARENTERAL NUTRITION IN NEWBORNS REQUIRING PROLONGED PARENTERAL NUTRITION
Brief Title: Impact of Cyclic Prolonged Parenteral Nutrition in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Manuel Sanchez Luna, Clinical Professor, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-12
Record Dates: First submitted 2015-12-16; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Cholestasis in Newborn
Keywords: intrahepatic cholestasis; infant newborn; cyclic parenteral nutrition
MeSH Terms: conditions — Cholestasis, Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Cyclic parenteral nutrition Cohort (Experimental): All newborn who were included in the study to receive cyclic parenteral nutrition (within 24 hours). The parenteral nutrition was stopped for one hour the first day until 4 hours in preterm infants and 6 hours in term neonates.
  Interventions: Procedure: Cyclic parenteral nutrition
- Control: Continuous parenteral nutrition (No Intervention): All newborn who were included in the study to receive continuous parenteral nutrition (24 hours). The parenteral nutrition was given by a central line in 24 hours with a basal flow

INTERVENTIONS:
Procedure: Cyclic parenteral nutrition — Cyclic parenteral nutrition was provided according to a method described by Longhurst et al. Patients were initially cycled of PN for 1 hour per day with increased rate of 1 hour with a maximum time out of PN of 4 hours for preterm babies < 37 weeks GA and 6 hours for term newborns. Glucose was monitored at half the time without PN to detect the hypoglycemia.
  Arms: Intervention: Cyclic parenteral nutrition Cohort

SUMMARY:
The aim of our study is to compare the incidence of PNAC in newborns receiving cyclic versus continuous parenteral nutrition (PN) in those newborns who need prolonged PN. The secondary aims are to compare incidence of sepsis and catheter related sepsis, mean length of hospital stay, mortality, nutritional status at two years of chronological age and predisposing factors to the development of parenteral nutrition associated cholestasis (PNAC) between the two groups, and to evaluate the adverse effects of the method of cycling used.

This was a single-center, prospective randomized not blinded study was conducted in a level 3 neonatal intensive care unit from July 2010 to January 2015. Infants with hemodynamic instability until a stable situation, congenital hepatic disease, preterm infants with diagnosis of respiratory distress syndrome or persistent ductus arteriosus and lack of authorization from the parents or guardians were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Newborns who needed long-term PN for more than ten days and were diagnosed with a pathology that makes likely the need to extend it.

Exclusion Criteria:

* Infants with hemodynamic instability until a stable situation, congenital hepatic disease, preterm infants with diagnosis of respiratory distress syndrome or persistent ductus arteriosus and lack of authorization from the parents or guardians

Ages: 10 Days to 50 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
% patients with parenteral nutrition associated cholestasis (PNAC) | through study completion, an average of 1 year
  The incidence of parenteral nutrition associated cholestasis in newborns receiving cyclic versus continuous PN in those newborns who need prolonged PN.

SECONDARY OUTCOMES:
Incidence of sepsis | through study completion, an average of 1 year
  The percentage of patients who was diagnosed of sepsis in newborns receiving cyclic versus continuous PN in those newborns who need prolonged PN.
Incidence of catheter related sepsis (CRS) | through study completion, an average of 1 year
  The percentage of patients who was diagnosed of CRS in newborns receiving cyclic versus continuous PN in those newborns who need prolonged PN.
Mean length of hospital stay | through study completion, an average of 1 year
  The mean length of hospital stay in newborns receiving cyclic versus continuous PN in those newborns who need prolonged PN.
Nutrition factors to the development of PNAC | through study completion, an average of 1 year
  total days on enteral nutrition in newborns receiving cyclic versus continuous PN in those newborns who need prolonged PN.
Nutrition factors to the development of PNAC | through study completion, an average of 1 year
  total days on parenteral nutrition in newborns receiving cyclic versus continuous PN in those newborns who need prolonged PN.
Anticholestatic drugs | through study completion, an average of 1 year
  % of patients with anticholestatic drug in newborns receiving cyclic versus continuous PN in those newborns who need prolonged PN.
Anticholestatic drugs | through study completion, an average of 1 year
  days of duration of treatment with anticholestatic drug in newborns receiving cyclic versus continuous PN in those newborns who need prolonged PN.
Adverse effects of the method of cycling used | through study completion, an average of 1 year
  Percentage of adverse effects, type of adverse affects
Mortality | through study completion, an average of 1 year
  the percentage of patients who died and the cause of death
Mortality | through study completion, an average of 1 year
  The cause of death

CONTACTS AND LOCATIONS:
Locations (1):
- Nelia Navarro patiño, Madrid, Madrid, Spain

REFERENCES:
- [Background] Angelico M, Della Guardia P. Review article: hepatobiliary complications associated with total parenteral nutrition. Aliment Pharmacol Ther. 2000 May;14 Suppl 2:54-7. doi: 10.1046/j.1365-2036.2000.014s2054.x. PMID 10903005